CLINICAL TRIAL: NCT06836297
Title: Neural and Behavioural Bases of Action Simulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NBBAS
Record Dates: First submitted 2025-02-10; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transcranial Magnetic Stimulation (Experimental): For some experiments, all participants will take part in all experimental conditions. For other experiments, participants will be randomly assigned to different groups with different conditions (e.g. TMS sham vs. TMS test).
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation Sham — Participants will be asked to perform various behavioral tasks involving the use of action observation or motor imagery. During these tasks, transcranial magnetic stimulation will be used.

SUMMARY:
The goal of this interventional study is to understand the neural and behavioural bases of action simulation and its links with action execution in healthy volunteers.

Hypotheses: Action simulation recruits neural networks that are largely similar to those activated by action execution, with some differences to avoid executing a movement while observing/imagining it.

Participants will be tested with TMS while doing motor imagery or action observation.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult volunteers (more than 18 years old)

Exclusion Criteria:

* Participants taking anti-epileptic drugs
* pregnant or breastfeeding women cannot participate in this study
* people with a pacemaker
* people with a cochlear implant
* people with a metal part in the brain or any other medical implant in their body (pump, neurostimulator, valve,) cannot take part in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Motor Evoked Potential (MEP) | For the duration of the participants' visit to the laboratory (max 2h30)
  Evoked motor potentials will be measured throughout the experiment using surface electrodes on different muscles to measure changes in corticospinal excitability.

IPD SHARING:
Plan to Share IPD: No